CLINICAL TRIAL: NCT01926314
Title: The Effect of Postpartum Pelvic Floor Rehabilitation in Prevention and Treatment of Pelvic Floor Dysfunction- a Multiple Centers Cooperation Research.
Brief Title: The Effect of Postpartum Pelvic Floor Rehabilitation in Prevention and Treatment of Pelvic Floor Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: pumch-gyn-06
Record Dates: First submitted 2013-08-17; First posted 2013-08-20 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Primiparous Women With Singleton Baby at Term

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- device (Experimental): Patients in this group will be offered pelvic floor muscle rehabilitation program using PHENIX Neuromuscular Stimulation Therapy System device. The participants will start therapy once a week 42 days after delivery, and last 8 weeks.
  Interventions: Device: PHENIX Neuromuscular Stimulation Therapy System device
- usual home care without device (Active Comparator): Patients in this group will receive usual home care without device.
  Interventions: Other: usual home care without device

INTERVENTIONS:
Device: PHENIX Neuromuscular Stimulation Therapy System device
  Arms: device
Other: usual home care without device
  Arms: usual home care without device

SUMMARY:
Pregnancy and childbirth are considered as risk periods for injuries to the pelvic floor and development of pelvic floor dysfunction. This may leed to devastating loss of function and quality of life.The aim of this study is to evaluate the effect of postpartum pelvic floor muscle training with the device "PHENIX Neuromuscular Stimulation Therapy Systems" on the recovery of pelvic floor function for primiparous women.

ELIGIBILITY:
Inclusion Criteria:

* primiparous delivery
* term delivery
* single childbirth
* aged from 18-50yrs

Exclusion Criteria:

* urinary incontinence before pregnancy
* fecal incontinence before pregnancy
* organ prolapse before pregnancy
* history of childbirth or induced labor with pregnancy more than 28 weeks
* multiparity
* newborn weight less than 2500 grams or more than 4000 grams
* precipitate labor
* complication of pregnancy
* asthma
* long-term abdominal pressure(chronic cough>1 month,chronic constipation)
* diabetes
* sciatica
* history of pelvic operation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2013-08; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
strength of deep muscle fiber I | 42 days after delivery
  Strength of deep muscle fiber I is one of the index of electrophysiology function of pelvic floor.
strength of deep muscle fiber I | 6 months after delivery
  Strength of deep muscle fiber I is one of the index of electrophysiology function of pelvic floor.
strength of deep muscle fiber I | 12 months after delivery
  Strength of deep muscle fiber I is one of the index of electrophysiology function of pelvic floor.
strength of deep muscle fiber II | 42 days after delivery
  Strength of deep muscle fiber II is one of the index of electrophysiology function of pelvic floor.
strength of deep muscle fiber II | 6 months after delivery
  Strength of deep muscle fiber II is one of the index of electrophysiology function of pelvic floor.
strength of deep muscle fiber II | 12 months after delivery
  Strength of deep muscle fiber II is one of the index of electrophysiology function of pelvic floor.
muscular fatigue level | 42 days after delivery
  muscular fatigue level is one of the index of electrophysiology function of pelvic floor.
muscular fatigue level | 6 months after delivery
  muscular fatigue level is one of the index of electrophysiology function of pelvic floor.
muscular fatigue level | 12 months after delivery
  muscular fatigue level is one of the index of electrophysiology function of pelvic floor.
myoelectric potential | 42 days after delivery
  myoelectric potential is one of the index of electrophysiology function of pelvic floor.
myoelectric potential | 6 months after delivery
  myoelectric potential is one of the index of electrophysiology function of pelvic floor.
myoelectric potential | 12 months after delivery
  myoelectric potential is one of the index of electrophysiology function of pelvic floor.
A3 reflex | 42 days after delivery
  A3 reflex is one of the index of urinary continence function of pelvic floor.
A3 reflex | 6 months after delivery
  A3 reflex is one of the index of urinary continence function of pelvic floor.
A3 reflex | 12 months after delivery
  A3 reflex is one of the index of urinary continence function of pelvic floor.
dynamic pressure of pelvic floor | 42 days after delivery
  dynamic pressure of pelvic floor is one of the index of urinary continence function.
dynamic pressure of pelvic floor | 6 months after delivery
  dynamic pressure of pelvic floor is one of the index of urinary continence function.
dynamic pressure of pelvic floor | 12 months after delivery
  dynamic pressure of pelvic floor is one of the index of urinary continence function.

SECONDARY OUTCOMES:
change from baseline in PFIQ-7 scores | 42 days after delivery
change from baseline in PFIQ-7 scores | 6 months after delivery
change from baseline in PFIQ-7 scores | 12 months after delivery
in subjects sexually active at baseline, assessment of sexual function using PISQ-12 | 42 days after delivery
in subjects sexually active at baseline, assessment of sexual function using PISQ-12 | 6 months after delivery
in subjects sexually active at baseline, assessment of sexual function using PISQ-12 | 12 months after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, Principal Investigator — Peking Union Medical College Hospital
Locations (4):
- China (4):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Foshan maternal and child health hospital, Foshan, Guangdong
  - The first affiliated hospital of Guangzhou medical college, Guangzhou, Guangdong
  - Wuxi Maternal and Child Health Hospital, Nanjing Medical University, Wuxi, Jiangsu